CLINICAL TRIAL: NCT00377195
Title: A Prospective Single Arm Trial of Involved Field Radiotherapy Alone for Stage I-II Low Grade Non-gastric Marginal Zone Lymphoma
Brief Title: Involved Field Radiotherapy for Non-gastric Marginal Zone Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Australasian Leukaemia and Lymphoma Group (Other); Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 05.02
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Non-gastric Marginal Zone Lymphoma
Keywords: Marginal Zone Lymphoma; Involved field radiotherapy; H. pylori
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Radiation: Involved Field Radiotherapy

INTERVENTIONS:
Radiation: Involved Field Radiotherapy — The prescribed dose will be 30 Gy in 15-20 fractions, unless the orbit is to be treated, in which case the dose will be 24 Gy in 1.5 to 2 Gy fractions.
  Daily fractions of 1.5-2.0 Gy will be employed. Treatment will be given 5 days per week with the planned duration of treatment not exceeding 28 days.
  Other Names: Radiation

SUMMARY:
This prospective study will test the following hypotheses in patients with stage I-II low grade marginal zone (MZ) lymphoma:

* Involved Field Radiotherapy will produce a complete response rate of > 90%
* Radiotherapy will be associated with a locoregional progression of < 20% after 10 years
* Death from MZ lymphoma will occur in < 40% of patients within 10 years of radiotherapy

This study secondary objectives are:

* To collect information on the prevalence of H. pylori in non-gastric MALT lymphoma
* To estimate rates of acute and late toxicity of radiotherapy

DETAILED DESCRIPTION:
Aims of the study :

* To conduct the first multicentre prospective trial of radiotherapy (RT) in stage I-II Marginal Zone Lymphoma (MZL)
* To prospectively identify causal factors for MZL, including infection and inflammatory disease

This study will be the first large trial of any form of therapy for stage I-II, non-gastric marginal zone lymphoma. There is an enormous deficit in the literature with respect to this fascinating but relatively recently-recognised entity. MZL is commonly associated with underlying inflammatory or infective disorders and it is clear, at least in some cases with infection by organisms called Helicobacter pylori and Chlamydia psitacci, that the inflammatory condition can actually cause the lymphoma. The role of H. pylori infection has not been well studied in non gastric MZL in large prospective studies, despite anecdotal reports of regression of non gastric MZL after H. pylori eradication. There have been reports of responses to doxycycline (antibacterial) therapy in patients with evidence of chlamydial infection (C. psitacci) in MZL of the tissues around the eye. This association has not been well studied in any large prospective study and no long-term data for doxycycline therapy exist. Management of stage I-II MZL is variable and often ad-hoc in Australia, despite significant retrospective evidence to support radiotherapy (RT) as the curative treatment modality of choice. In this TROG/ALLG joint study, 100 patients will be recruited over 5 years. All patients will undergo breath tests or endoscopy to detect H. pylori infection. Ocular MZL specimens will be sent to Italy to test for C. psitacci. Patients will receive highly standardised treatment with RT. This study will definitively document the efficacy and safety of RT in stage I and II non-gastric MZL and will include patients with stage IV disease limited to paired-organs, as this disease shows a tendency to home in exclusively on particular organs, such as salivary glands.

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years old with histologically documented non-gastric marginal zone lymphoma.
* Disease limited to stages I and II after adequate staging (see Appendix II), patients with stage IV with extranodal disease confined to paired organs (e.g. salivary glands) and including any local extension of this disease into adjacent tissues. Patients with involved lymph nodes on the same side of the diaphragm in addition to paired organ involvement are also eligible, provided all involved tumour sites, nodal and extranodal, can be irradiated to 30 Gy within the tolerance of the relevant normal tissues. If paired organ involvement was regarded as a single extranodal site (rather than 2 separate sites and hence stage IV), eligible patients would then be regarded as having stage IE or IIE disease. Patients with wider dissemination (bone marrow, liver etc) are ineligible.
* Anticipated life expectancy > 2 years
* Given written informed consent
* Been assessed by a radiation oncologist
* Agree to undergo breath testing for H. pylori and/or oesophagogastroduodenoscopy to exclude active infection with helicobacter pylori
* Must be available for long-term follow up

Exclusion Criteria:

* Splenic marginal zone lymphoma
* Received previous locoregional radiotherapy
* A medical contraindication to radiotherapy
* Any previous or concurrent malignancy other than curatively treated non-melanoma skin cancer, level 1 malignant melanoma, or in situ cervical cancer, unless disease and treatment-free for 5 years
* Such extensive involvement of the thorax that treatment with radiotherapy alone would be hazardous because of excessive lung irradiation, even if a shrinking field technique were employed
* Suspected or confirmed pregnancy
* Transformation to large cell lymphoma or other aggressive histology
* Disease that is widely disseminated (bone marrow, liver etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-07-08 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Freedom from locoregional progression (FFLRP) rate | There will be an interim analysis at the end of accual (approx 5 years), at 5 years from the end of accrual and a final analysis at 10 years form the end of accrual.
Complete response rate | A final analysis at 10 years form the end of accrual.
Cancer-specific survival | A final analysis at 10 years form the end of accrual.

SECONDARY OUTCOMES:
Overall survival | A final analysis at 10 years form the end of accrual.
Progression free survival | A final analysis at 10 years form the end of accrual.
Freedom from progression | A final analysis at 10 years form the end of accrual.
Acute and Late Toxicity rates | There will be an interim analysis at the end of accual (approx 5 years), at 5 years from the end of accrual and a final analysis at 10 years form the end of accrual.

CONTACTS AND LOCATIONS:
Overall Officials: Michael MacManus, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (5):
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

REFERENCES:
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au